CLINICAL TRIAL: NCT05885737
Title: A Randomised, Double-Blind, Placebo-Controlled, Multicentre, Phase 3, Clinical Study of Difelikefalin in Haemodialysis Chinese Adult Subjects With Moderate-to-Severe Pruritus
Brief Title: Phase 3 Study of Difelikefalin in Haemodialysis Chinese Adult Subjects With Moderate-to-Severe Pruritus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vifor Fresenius Medical Care Renal Pharma (Industry)
Collaborators: Tigermed Consulting Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KOR-CHINA-301; CTR20220844 (Other: China CTR Number)
Record Dates: First submitted 2023-05-17; First posted 2023-06-02 (Actual); Results first posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Uremic Pruritus
Keywords: Uremic Pruritus; Chronic kidney disease-associated pruritus; CKD-aP; Difelikefalin
MeSH Terms: interventions — difelikefalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 12-weeks double-blind period - Difelikefalin (Experimental)
  Interventions: Drug: Difelikefalin Injection
- 12-weeks double-blind period - Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Injection
- 14-weeks optional open-label period following the double-blind period - Difelikefalin (Experimental)
  Interventions: Drug: Difelikefalin Injection

INTERVENTIONS:
Drug: Difelikefalin Injection — Participants receive Difelikefalin three times a week (0.5 micrograms/kg dry body weight). Difelikefalin is administered by intravenous bolus injection into the venous line of the dialysis circuit at the end of each dialysis.
  Arms: 12-weeks double-blind period - Difelikefalin; 14-weeks optional open-label period following the double-blind period - Difelikefalin
Drug: Placebo Injection — Participants receive Placebo three times a week (0.5 micrograms/kg dry body weight). Placebo is administered by intravenous bolus injection into the venous line of the dialysis circuit at the end of each dialysis.
  Arms: 12-weeks double-blind period - Placebo

SUMMARY:
This a multicentre study that consists of a 12-week double-blind period, and an optional 14-week open-label extension period and a 1-week follow-up period.

DETAILED DESCRIPTION:
Total study duration for a single subject is 31 to 32 weeks with a 4-week screening period, a 12-week double-blind period, a 14-week optional open-label extension period, and a 1-week follow-up period. For subjects not participating in the open-label extension period, the total study duration is 17 weeks.

Difelikefalin will be administered in the double-blind and open-label period 3 times a week at the end of each dialysis session. The total dose of the investigational product will be determined based on the subject's prescription dry body weight.

The primary objective of the study is:

To evaluate the efficacy of difelikefalin 0.5 μg/kg compared to placebo in reducing the intensity of itch in HD Chinese subjects with moderate-to-severe pruritus.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with chronic kidney disease (CKD) on HD 3 times weekly for ≥12 weeks prior to the informed consent procedure (including the date of informed consent) who can continue HD without changing its frequency or method.
* If female, is not pregnant, or nursing.
* If female:

  1. Is surgically sterile; or
  2. Has been amenorrhoeic for at least 1 year and is over the age of 55 years; or
  3. Has a negative serum pregnancy test within 7 days before first dose of investigational product and agrees to use acceptable contraceptive measures (e.g., hormonal contraceptives, barrier with spermicide, intrauterine device, vasectomised partner, or abstinence) from the time of informed consent until 7 days after the last dose of investigational product.
* If male, agrees not to donate sperm after the first dose of investigational product administration until 7 days after the last dose of investigational product, and agrees to use a condom with spermicide or abstain from heterosexual intercourse during the study until 7 days after the last dose of investigational product.
* Subjects with a prescription dry body weight between 40 and 100 kg, inclusive.

Exclusion Criteria:

* Planned or anticipated to receive a kidney transplant during the study.
* Has localised itch restricted to the palms of the hands.
* Has pruritus only during the dialysis session
* Subjects with severe hepatic impairment (Child-Pugh Class C) or concurrent hepatic cirrhosis.
* Subject is receiving ongoing ultraviolet B treatment and anticipates receiving such treatment during the study.
* Significant systolic or diastolic heart failure (e.g., New York Heart Association Class IV congestive heart failure)
* Subjects with concurrent malignancy except excised basal cell or squamous cell carcinoma of the skin, or carcinoma in situ that has been excised or resected completely.
* Known or suspected history of alcohol, narcotic, or other drug abuse, or substance dependence within 12 months prior to screening.
* Severe mental illness or cognitive impairment (e.g., dementia) or other concurrent mental disorder that, in the opinion of the Investigator, would compromise the validity of study measurements.
* Any other relevant acute or chronic medical or neuropsychiatric condition within 3 months prior to screening (e.g., diagnosis of encephalopathy, coma, delirium).
* New or change of treatment received for itch including antihistamines and corticosteroids (oral, IV, or topical) within 14 days prior to screening.
* New or change of prescription for opioids, gabapentin, or pregabalin within 14 days prior to screening.
* Subject is receiving prohibited medication (e.g., nalfurafine hydrochloride, opioid antagonists)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2023-05-18 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Milica Enoiu, PhD, Study Director — Vifor Pharma Group
Locations (35):
- China (35):
  - Investigator Site 25, Baotou
  - Investigator Site 01, Beijing
  - Investigator Site 07, Beijing
  - Investigator Site 26, Changsha
  - Investigator Site 06, Guangzhou
  - Investigator Site 12, Jiaxing
  - Investigator Site 02, Lanzhou
  - Investigator Site 34, Mianyang
  - Investigator Site 03, Nanjing
  - Investigator Site 10, Nanjing
  - Investigator Site 19, Nanjing
  - Investigator Site 36, Nantong
  - Investigator Site 40, Shanghai
  - Investigator Site 18, Shenyang
  - Investigator Site 21, Shenyang
  - Investigator Site 16, Shenzhen
  - Investigator Site 08, Shihezi
  - Investigator Site 32, Shijiazhuang
  - Investigator Site 41, Shijiazhuang
  - Investigator Site 20, Taiyuan
  - Investigator Site 24, Taiyuan
  - Investigator Site 39, Tianjin
  - Investigator Site 04, Ürümqi
  - Investigator Site 17, Wuhan
  - Investigator Site 33, Wuxi
  - Investigator Site 13, Xiamen
  - Investigator Site 15, Xianyang
  - Investigator Site 22, Xining
  - Investigator Site 38, Xinxiang
  - Investigator Site 11, Yangzhou
  - Investigator Site 30, Yibin
  - Investigator Site 29, Yinchuan
  - Investigator Site 23, Zhengzhou
  - Investigator Site 31, Zhenjiang
  - Investigator Site 35, Zhuzhou

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider on a case-by-case basis requests to share Individual Patient Data (IPD) with external bona-fide, qualified scientific and medical researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
Time Frame: Requests for IPD will generally be considered once review by major regulatory authorities (ie FDA, EMA) is complete and the primary publication is available.
Access Criteria: Proposed research should seek to answer a previously unanswered important medical or scientific question.
  Applicable country-specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 35 investigative sites in China.
Pre-assignment Details: A total of 291 participants were screened, and 31 of these were screen failures. Of the screened participants, 260 were randomized in the study. Of these 260 participants, 227 completed the double blind (DB) treatment period and 217 of these participants entered the open-label extension (OLE) period of the study.
Groups:
- Difelikefalin/Difelikefalin: Participants received Difelikefalin injected into the venous line of the dialysis circuit at the end of each dialysis session for up to 12 weeks (3 times weekly, 36 times in total) in the DB period. Upon completion of the DB period, participants who chose to enter the optional OLE period received Difelikefalin additionally for up to 14 weeks (3 times weekly), starting at Week 13, and until Week 26 inclusive.
- Placebo/Difelikefalin: Participants received Placebo injected into the venous line of the dialysis circuit at the end of each dialysis session matching to Difelikefalin for up to 12 weeks (3 times weekly, 36 times in total) in the DB period. Upon completion of the DB period, participants who chose to enter the optional OLE period received Difelikefalin additionally for up to 14 weeks (3 times weekly), starting at Week 13, and until Week 26 inclusive.
Period: DB Period
Arm/Group | Difelikefalin/Difelikefalin | Placebo/Difelikefalin
Started | 130 | 130
Treated | 129 | 130
Completed | 110 | 117
Not Completed | 20 | 13
Not completed — Adverse Event | 4 | 4
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 12 | 6
Not completed — Other: Unspecified | 2 | 2
Period: OLE Period
Arm/Group | Difelikefalin/Difelikefalin | Placebo/Difelikefalin
Started | 103 (Participants who entered the OLE period upon completion of DB period.) | 114 (Participants who entered the OLE period upon completion of DB period.)
Treated | 103 | 113
Completed | 92 | 106
Not Completed | 11 | 8
Not completed — Adverse Event | 3 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 5 | 5
Not completed — Other: Unspecified | 2 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on the full analysis set (FAS). The FAS included all participants who were randomised to treatment, received at least 1 dose of investigational product and had a non-missing baseline assessment for the weekly mean of the daily 24-hour Worst Itch Numeric Rating Scale (WI-NRS) score.
Groups:
- DB Period: Difelikefalin: Participants received Difelikefalin injected into the venous line of the dialysis circuit at the end of each dialysis session for up to 12 weeks (3 times weekly, 36 times in total).
- DB Period: Placebo: Participants received Placebo injected into the venous line of the dialysis circuit at the end of each dialysis session matching to Difelikefalin for up to 12 weeks (3 times weekly, 36 times in total).
- Total: Total of all reporting groups
Arm/Group | DB Period: Difelikefalin | DB Period: Placebo | Total
Number analyzed (Participants) | 129 | 130 | 259
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (12.26) | 55.7 (12.38) | 56.0 (12.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 42 | 86
  Male | 85 | 88 | 173
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - Chinese | 129 | 130 | 259
WI-NRS [Mean (Standard Deviation); unit: score on a scale] | 7.35 (1.291) | 7.00 (1.223) | 7.18 (1.268)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Weekly Mean of the Daily 24-hour WI-NRS Score at Week 4 of the DB Period
Description: On a daily basis, participants recorded the intensity of the worst itching they experienced over the past 24 hours using a numerical rating scale (NRS) scale from 0 to 10, where 0 represents "no itching" and 10 was "worst itching imaginable". A higher score indicated a more severe outcome. The weekly mean of the daily values of the daily 24-hour WI-NRS was calculated for the analysis. The least square (LS) means of change from baseline to Week 4 in the weekly mean of the daily 24-hour WI-NRS score was estimated using the mixed model repeated measures (MMRM) method. The MMRM model included use of prior anti-itch medication (yes/no), presence of specific medical conditions at baseline (yes/no), treatment, visit, and treatment-by-visit-interaction as fixed categorical effects and baseline WI-NRS score as fixed continuous effects.
Time Frame: From Baseline to Week 4
Population: Analysis was performed on the FAS. The FAS included all participants who were randomized to treatment, received at least 1 dose of investigational product and had a non-missing baseline assessment for the weekly mean of the daily 24-hour WI-NRS score. Here, 'overall number of participants analyzed', 'N' = participants with available data for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | DB Period: Difelikefalin | DB Period: Placebo
Number analyzed (Participants) | 119 | 126
score on a scale | -2.09 (0.198) | -1.27 (0.194)
Statistical Analysis 1: Comparison: DB Period: Difelikefalin vs DB Period: Placebo; The null hypothesis in this study was that there was no treatment difference in the primary efficacy analysis of the primary endpoint. The alternative hypothesis was that in participants randomized to difelikefalin there was a significant treatment difference in change in itching compared to participants randomized to placebo. The assessment was based on the mean change from baseline in the weekly mean of the daily 24-hour WI-NRS score at Week 4 of the DB period; Test type: Equivalence — Testing of primary efficacy endpoint was 2-sided and conducted at the 5% significance level. The efficacy of difelikefalin was to be declared for this study if null hypothesis of no treatment difference in the primary efficacy analysis was rejected in favor of the alternative that participants randomized to difelikefalin experience significantly different itching compared to participants randomized to placebo. The null hypothesis was to be rejected if the 2-sided p value was less than (<) 0.05; p = 0.0003, MMRM; Least square mean difference = -0.81, 95% CI 2-sided [-1.25 to -0.37], Standard Error of Mean 0.223

2. Secondary Outcome: Percentage of Participants Achieving Greater Than or Equal to (>=) 3-point Improvement From Baseline With Respect to the Weekly Mean of the Daily 24-hour WI-NRS in the DB Period
Description: On a daily basis, participants recorded the intensity of the worst itching they experienced over the past 24 hours using a NRS scale from 0 to 10, where 0 represents "no itching" and 10 was "worst itching imaginable". A higher score indicated a more severe outcome. The weekly mean of the daily values of the daily 24-hour WI-NRS was calculated for the analysis. Missing weekly mean WI-NRS data were imputed using missing at random (MAR) multiple imputation (MI) approach, assuming that participants who do not have weekly mean WI-NRS score at a timepoint would have similar weekly mean WI-NRS scores as other participants in their respective treatment arm who have complete data. The percentage of participants were estimated using a logistic regression model with terms for treatment group, baseline WI-NRS score, use of anti-itch medication during the week prior to randomisation, and the presence of specific medical conditions at baseline.
Time Frame: From Baseline, and at Weeks 4, 8, and 12
Population: Analysis was performed on FAS. The FAS included all participants who were randomized to treatment, received at least 1 dose of investigational product and had a non-missing baseline assessment for the weekly mean of the daily 24-hour WI-NRS score. Here, 'number analyzed', 'n' = participants with available data for each specified timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | DB Period: Difelikefalin | DB Period: Placebo
Number analyzed (Participants) | 129 | 130
percentage of participants
  Week 4: number analyzed (Participants) | 119 | 126
  Week 4 | 21.9 [11.4 to 38.1] | 8.9 [3.9 to 19.0]
  Week 8: number analyzed (Participants) | 114 | 121
  Week 8 | 35.8 [22.7 to 51.3] | 22.3 [12.9 to 35.8]
  Week 12: number analyzed (Participants) | 110 | 119
  Week 12 | 48.7 [34.2 to 63.3] | 33.8 [22.0 to 48.0]

3. Secondary Outcome: Percentage of Participants Achieving at Least 4-point Improvement From Baseline With Respect to the Weekly Mean of the Daily 24-hour WI-NRS in the DB Period
Description: On a daily basis, participants recorded the intensity of the worst itching they experienced over the past 24 hours using a NRS scale from 0 to 10, where 0 represents "no itching" and 10 was "worst itching imaginable". A higher score indicated a more severe outcome. The weekly mean of the daily values of the daily 24-hour WI-NRS was calculated for the analysis. Missing weekly mean WI-NRS data were imputed using MAR-MI approach, assuming that participants who do not have weekly mean WI-NRS score at a timepoint would have similar weekly mean WI-NRS scores as other participants in their respective treatment arm who have complete data.
Time Frame: From Baseline, and at Weeks 4, 8, and 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | DB Period: Difelikefalin | DB Period: Placebo
Number analyzed (Participants) | 129 | 130
percentage of participants
  Week 4: number analyzed (Participants) | 119 | 126
  Week 4 | 10.9 [3.7 to 28.1] | 2.2 [0.5 to 8.8]
  Week 8: number analyzed (Participants) | 114 | 121
  Week 8 | 21.2 [11.2 to 36.6] | 11.6 [5.4 to 23.2]
  Week 12: number analyzed (Participants) | 110 | 119
  Week 12 | 29.9 [18.1 to 45.3] | 19.7 [10.9 to 32.9]

4. Secondary Outcome: Change From Baseline in the Weekly Mean of the 24-hour WI-NRS Score at Each Week of the DB Period
Description: On a daily basis, participants recorded the intensity of the worst itching they experienced over the past 24 hours using a NRS scale from 0 to 10, where 0 represents "no itching" and 10 was "worst itching imaginable". A higher score indicated a more severe outcome. The weekly mean of the daily values was calculated for the analysis. The weekly mean of the daily values of the daily 24-hour WI-NRS was calculated for the analysis. The MMRM model included use of prior anti-itch medication (yes/no), presence of specific medical conditions at baseline (yes/no), treatment, visit, and treatment-by-visit-interaction as fixed categorical effects and baseline WI-NRS score as fixed continuous effects.
Time Frame: From Baseline to Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | DB Period: Difelikefalin | DB Period: Placebo
Number analyzed (Participants) | 129 | 130
score on a scale
  Week 1: number analyzed (Participants) | 128 | 130
  Week 1 | -0.68 (0.153) | -0.53 (0.149)
  Week 2: number analyzed (Participants) | 126 | 128
  Week 2 | -1.37 (0.179) | -0.89 (0.175)
  Week 3: number analyzed (Participants) | 122 | 126
  Week 3 | -1.86 (0.188) | -1.08 (0.185)
  Week 4: number analyzed (Participants) | 119 | 126
  Week 4 | -2.09 (0.198) | -1.27 (0.194)
  Week 5: number analyzed (Participants) | 117 | 123
  Week 5 | -2.35 (0.208) | -1.46 (0.204)
  Week 6: number analyzed (Participants) | 118 | 123
  Week 6 | -2.51 (0.216) | -1.55 (0.212)
  Week 7: number analyzed (Participants) | 115 | 121
  Week 7 | -2.61 (0.219) | -1.78 (0.215)
  Week 8: number analyzed (Participants) | 114 | 121
  Week 8 | -2.71 (0.222) | -1.96 (0.217)
  Week 9: number analyzed (Participants) | 114 | 120
  Week 9 | -2.90 (0.223) | -2.00 (0.218)
  Week 10: number analyzed (Participants) | 113 | 120
  Week 10 | -2.97 (0.227) | -2.04 (0.222)
  Week 11: number analyzed (Participants) | 111 | 120
  Week 11 | -3.08 (0.228) | -2.16 (0.223)
  Week 12: number analyzed (Participants) | 110 | 119
  Week 12 | -3.11 (0.235) | -2.16 (0.229)

5. Secondary Outcome: Change From Baseline in Itch-related Quality-of-life (QoL) as Assessed by the 5-D Itch Scale Total Score (DB Period)
Description: The 5-D itch scale is a questionnaire where participants assess the 5 dimensions of itch (degree, duration, direction, disability, and distribution). The scores of each of the 5 domains are achieved separately and then summed together to obtain a total 5-D score. 5-D itch scale scores can potentially range between 5 (no pruritus) and 25 (most severe pruritus) where a higher score indicates a more severe outcome. The LS means of change from baseline in itch-related QoL as assessed by the 5-D itch scale total score was estimated using the MMRM method. The MMRM model included use of prior anti-itch medication (yes/no), presence of specific medical conditions at baseline (yes/no), treatment sequence, visit, and treatment sequence-by-visit-interaction as fixed categorical effects and baseline 5-D Itch score (total score) as fixed continuous effects.
Time Frame: From Baseline to Weeks 4, 8, and 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | DB Period: Difelikefalin | DB Period: Placebo
Number analyzed (Participants) | 129 | 130
score on a scale
  Week 4: number analyzed (Participants) | 119 | 125
  Week 4 | -3.3 (0.37) | -2.5 (0.36)
  Week 8: number analyzed (Participants) | 114 | 121
  Week 8 | -3.9 (0.38) | -2.8 (0.37)
  Week 12: number analyzed (Participants) | 111 | 119
  Week 12 | -4.3 (0.40) | -3.6 (0.39)

6. Secondary Outcome: Change From Baseline in Itch-related QoL as Assessed by the 5-D Itch Scale Total Score (OLE Period)
Description: as for outcome 5
Time Frame: From Baseline to OLE Period - Weeks 4, 8, 12, and 14
Population: Analysis was performed on the OLE Safety Analysis Set, which included all participants who received at least 1 dose of IP in the OLE period. Here, 'number analyzed', 'n' = participants with available data for each specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- OLE Period: Difelikefalin/Difelikefalin: Upon completion of the DB period, participants who received Difelikefalin in DB period, who chose to enter the optional OLE period, received Difelikefalin additionally for up to 14 weeks (3 times weekly), starting at Week 13, and until Week 26 inclusive.
- OLE Period: Placebo/Difelikefalin: Upon completion of the DB period, participants who received placebo in DB period, who chose to enter the optional OLE period, received Difelikefalin additionally for up to 14 weeks (3 times weekly), starting at Week 13, and until Week 26 inclusive.
Arm/Group | OLE Period: Difelikefalin/Difelikefalin | OLE Period: Placebo/Difelikefalin
Number analyzed (Participants) | 103 | 113
score on a scale
  Week 4: number analyzed (Participants) | 97 | 107
  Week 4 | -5.0 (0.40) | -5.3 (0.38)
  Week 8: number analyzed (Participants) | 92 | 105
  Week 8 | -5.4 (0.40) | -5.8 (0.37)
  Week 12: number analyzed (Participants) | 91 | 104
  Week 12 | -5.7 (0.41) | -6.0 (0.39)
  Week 14: number analyzed (Participants) | 90 | 101
  Week 14 | -6.2 (0.41) | -6.0 (0.38)

7. Secondary Outcome: Change From Baseline in Itch-related QoL as Assessed by the Skindex-10 Scale Total Score (DB Period)
Description: The Skindex-10 scale is a questionnaire that measures QoL in relationship to the itch intensity. Participants are asked the question "During the past week, how often have you been bothered by" and respond by filling in 1 of 7 circles numbered from 0 (labelled with the anchor phrase "never bothered") to 6 (labelled as "always bothered") for each of the 10 questions. The total score is the sum of the numeric value of each answered question. Here, a higher score indicated a severe outcome. The LS means of change from baseline in itch-related QoL as assessed by the Skindex-10 scale total score was estimated using the MMRM method. The MMRM model included use of prior anti-itch medication (yes/no), presence of specific medical conditions at baseline (yes/no), treatment, visit, and treatment-by-visit-interaction as fixed categorical effects and baseline skindex-10 scale score (total score) as fixed continuous effects.
Time Frame: From Baseline to Weeks 4, 8, and 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | DB Period: Difelikefalin | DB Period: Placebo
Number analyzed (Participants) | 129 | 130
score on a scale
  Week 4: number analyzed (Participants) | 120 | 124
  Week 4 | -9.1 (1.46) | -5.1 (1.43)
  Week 8: number analyzed (Participants) | 115 | 121
  Week 8 | -11.3 (1.51) | -7.4 (1.48)
  Week 12: number analyzed (Participants) | 111 | 119
  Week 12 | -10.5 (1.59) | -9.5 (1.55)

8. Secondary Outcome: Change From Baseline in Itch-related QoL as Assessed by the Skindex-10 Scale Total Score (OLE Period)
Description: as for outcome 7
Time Frame: From Baseline to OLE Period - Weeks 4, 8, 12, and 14
Population: For the OLE period analysis was performed on OLE-SAS, which included all participants who received at least 1 dose of IP in the OLE period. Here, 'number analyzed', 'n' = participants with available data for each specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | OLE Period: Difelikefalin/Difelikefalin | OLE Period: Placebo/Difelikefalin
Number analyzed (Participants) | 103 | 113
score on a scale
  Week 4: number analyzed (Participants) | 97 | 107
  Week 4 | -14.7 (1.47) | -14.1 (1.39)
  Week 8: number analyzed (Participants) | 93 | 106
  Week 8 | -15.8 (1.49) | -15.2 (1.41)
  Week 12: number analyzed (Participants) | 91 | 105
  Week 12 | -17.5 (1.48) | -16.4 (1.39)
  Week 14: number analyzed (Participants) | 91 | 102
  Week 14 | -18.3 (1.56) | -15.8 (1.48)

9. Secondary Outcome: Patient Global Impression of Change
Description: The Patient Global Impression of Change is a global participant reported outcome measure that assesses the change in itch (no change, improvement or worsening) overall relative to the start of the study. The scale has only 1 item, and the participant was asked to mark the category that best describes the change in itch ranging from "Very Much Improved" to "Very Much Worse". Number of participants within all individual categories are reported here.
Time Frame: At Week 12
Population: Analysis was performed on FAS. The FAS included all participants who were randomized to treatment, received at least 1 dose of investigational product and had a non-missing baseline assessment for the weekly mean of the daily 24-hour WI-NRS score. Here, 'overall number of participants analyzed', 'N' = participants with available data for the outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | DB Period: Difelikefalin | DB Period: Placebo
Number analyzed (Participants) | 110 | 119
Participants
  Very much improved | 20 | 14
  Much improved | 46 | 29
  Minimally improved | 22 | 49
  No change | 18 | 24
  Minimally worse | 2 | 2
  Much worse | 2 | 1
  Very Much worse | 0 | 0

10. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Time Frame: Up to Week 27 (12 weeks in DB + 14 weeks in OLE +1 week of follow up)
Population: Analysis was performed on safety analysis set in DB period (DB-SAF). DB-SAF included all randomized participants who received at least 1 dose of investigational product during the DB period. For the OLE period analysis was performed on OLE Safety Analysis Set, which included all participants who received at least 1 dose of IP in the OLE period.
Measure: Count of Participants; unit: Participants
Arm/Group | DB Period: Difelikefalin | DB Period: Placebo | OLE Period: Difelikefalin/Difelikefalin | OLE Period: Placebo/Difelikefalin
Number analyzed (Participants) | 129 | 130 | 103 | 113
Participants | 106 | 92 | 82 | 90

11. Secondary Outcome: Number of Participants With Clinically Significant Abnormal 12-lead Electrocardiogram (ECG)
Time Frame: Up to Week 27 (12 weeks in DB + 14 weeks in OLE +1 week of follow up)
Population: The DB and OLE SAS consisted of all participants who received at least 1 dose of investigational product during the DB period and OLE period, respectively. Participants were analysed according to the actual treatment received. Here, 'number analyzed', 'n' = participants with available data for each specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Difelikefalin/Difelikefalin | Placebo/Difelikefalin
Number analyzed (Participants) | 129 | 130
Participants
  DB period: Week 12: number analyzed (Participants) | 99 | 107
  DB period: Week 12 | 41 | 48
  OLE period: Week 14: number analyzed (Participants) | 84 | 100
  OLE period: Week 14 | 34 | 46

12. Secondary Outcome: Number of Participants With Clinically Relevant Change From Baseline in Vital Signs and Laboratory Evaluations
Time Frame: From baseline to Week 27 (12 weeks in DB + 14 weeks in OLE +1 week of follow up)
Population: The DB and OLE SAS consisted of all participants who received at least 1 dose of investigational product during the DB period and OLE period, respectively. Participants were analysed according to the actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Difelikefalin/Difelikefalin | Placebo/Difelikefalin
Number analyzed (Participants) | 129 | 130
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From Baseline up to Week 27 (12 weeks in DB + 14 weeks in OLE +1 week of follow-up)
Description: The DB and OLE SAS consisted of all participants who received at least 1 dose of investigational product during the DB period and OLE period, respectively. Participants were analysed according to the actual treatment received.
Groups:
- OLE Period: Difelikefalin/Difelikefalin: Upon completion of the double-blind period, participants who received Difelikefalin in DB period, who chose to enter the optional OLE period, received Difelikefalin additionally for up to 14 weeks (3 times weekly), starting at Week 13, and until Week 26 inclusive.
- OLE Period: Placebo/Difelikefalin: Upon completion of the double-blind period, participants who received placebo in DB period, who chose to enter the optional OLE period, received Difelikefalin additionally for up to 14 weeks (3 times weekly), starting at Week 13, and until Week 26 inclusive.
Arm/Group | DB Period: Difelikefalin | DB Period: Placebo | OLE Period: Difelikefalin/Difelikefalin | OLE Period: Placebo/Difelikefalin
All-Cause Mortality (participants affected / at risk) | 0/129 | 0/130 | 0/103 | 0/113
Serious Adverse Events (participants affected / at risk) | 18/129 | 12/130 | 19/103 | 12/113
Other Adverse Events (participants affected / at risk) | 85/129 | 66/130 | 65/103 | 69/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DB Period: Difelikefalin (N=129) | DB Period: Placebo (N=130) | OLE Period: Difelikefalin/Difelikefalin (N=103) | OLE Period: Placebo/Difelikefalin (N=113)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial injury (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Corneal opacity (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal artery occlusion (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract cortical (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Venous stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal cyst haemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular access placement (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DB Period: Difelikefalin (N=129) | DB Period: Placebo (N=130) | OLE Period: Difelikefalin/Difelikefalin (N=103) | OLE Period: Placebo/Difelikefalin (N=113)
Hyperkalaemia (Metabolism and nutrition disorders) | 21 (27) | 21 (25) | 20 (32) | 21 (34)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (3) | 7 (7) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 5 (5) | 6 (6)
Dialysis hypotension (Vascular disorders) | 19 (71) | 9 (26) | 13 (55) | 16 (63)
Hypotension (Vascular disorders) | 21 (29) | 8 (11) | 11 (12) | 15 (28)
Upper respiratory tract infection (Infections and infestations) | 13 (15) | 14 (16) | 9 (9) | 11 (14)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 18 (39) | 11 (15) | 11 (30) | 15 (33)
Tachycardia (Cardiac disorders) | 6 (16) | 6 (37) | 3 (4) | 9 (48)
Palpitations (Cardiac disorders) | 8 (10) | 5 (7) | 4 (4) | 7 (11)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 6 (6) | 7 (7) | 3 (3)
Constipation (Gastrointestinal disorders) | 9 (11) | 4 (4) | 4 (4) | 1 (3)
Dizziness (Nervous system disorders) | 16 (18) | 8 (16) | 6 (7) | 6 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 7 (8) | 6 (8) | 2 (2)
Insomnia (Psychiatric disorders) | 7 (10) | 4 (5) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2022-03-30): https://cdn.clinicaltrials.gov/large-docs/37/NCT05885737/Prot_000.pdf
  • Statistical Analysis Plan: DB Period (2024-08-12): https://cdn.clinicaltrials.gov/large-docs/37/NCT05885737/SAP_001.pdf
  • Statistical Analysis Plan: OLE Period (2024-11-28): https://cdn.clinicaltrials.gov/large-docs/37/NCT05885737/SAP_002.pdf